CLINICAL TRIAL: NCT07260916
Title: Minimally Invasive Neuroendoscopic Ultra-Early Targeted ICH Evacuation (MINUTE) Trial
Brief Title: Minimally Invasive Neuroendoscopic Ultra-Early Targeted ICH Evacuation
Acronym: MINUTE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Beth Israel Deaconess Medical Center (Other); Medical University of South Carolina (Other); NINDS Stroke Trials Network (StrokeNet) (Other)
Responsible Party: Principal Investigator, J. Mocco, National Principal Investigator, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GCO 23-1905; 1UG3NS138638-01A1 (NIH)
Record Dates: First submitted 2025-11-07; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Basal Ganglia Intracerebral Hemorrhage
Keywords: Basal Ganglia; SCUBA; Intracerebral Hemorrhage
MeSH Terms: conditions — Cerebral Hemorrhage

STUDY DESIGN:
Intervention Model Description: Adult patients (18-80 years old) with spontaneous Basal Ganglia (BG) intracerebral hemorrhage (ICH) ≥20 mL able to be randomized for endoscopic evacuation within 16 hours of ICH onset or last known well (LKW). Endoscopic minimally invasive Stereotactic Cerebral Underwater Blood Aspiration (SCUBA) of spontaneous basal ganglia ICH (BGH)
Who Masked: Outcomes Assessor
Masking Description: MINUTE is an on-label study with a blinded end-point outcome assessment, i.e. participants, providers, and site investigators will not be blinded to treatment assignments. Blinding is difficult, if not impossible, from a clinical perspective. It is not possible to blind the Investigator who treats the patient, the clinical staff, or the research team. Physicians treating participants who experience an AE after must know how the hemorrhage was treated in order to effectively report the AE and plan further treatment. However, MINUTE will require that study-related follow-up assessments be conducted by blinded investigators certified in mRS assessment, who were not involved in clinical care of the participant and are unaware of the patient's randomization status. A large Band-Aid will be placed on every patient's forehead prior to blinded assessor review, thereby preventing scar visualization or misinterpretation of unrelated scars on control patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Endoscopic ICH evacuation (SCUBA) and Standard Medical Treatment (Experimental): Participants will be treated with SCUBA and Standard Medical Treatment
  Interventions: Procedure: Endoscopic ICH evacuation; Other: Standard Medical Treatment
- Standard Medical Treatment (Placebo Comparator): Participants will be treated with Standard Medical Treatment
  Interventions: Other: Standard Medical Treatment

INTERVENTIONS:
Procedure: Endoscopic ICH evacuation — The intervention is minimally invasive endoscopic ICH evacuation using the SCUBA approach29. Stereotactic guidance must be used to guide placement of the sheath into the hematoma. Using stereotactic guidance software, a trajectory is planned along the long axis of the hematoma to the skull while avoiding eloquent brain regions, prominent vasculature, and other anatomy that should not be traversed during the approach, such as the frontal sinuses. A tele-proctor will be available to review the trajectory prior to the procedure starting. The procedure is performed under general anesthesia. The patient's head can be fixed if required depending on the stereotactic navigation system used.
  Other Names: SCUBA
  Arms: Endoscopic ICH evacuation (SCUBA) and Standard Medical Treatment
Other: Standard Medical Treatment — Participating physicians will attest that they will manage all ICH patients in the medical and surgical arms of the trial according to their institutional standards of care, which they will attest are consistent with the American Stroke Association guidelines for management of spontaneous ICH66 and utilize a standardized blood pressure management and hydrocephalus management protocol.

SUMMARY:
MINUTE is a prospective, multi-center, randomized, controlled, blinded assessor, adaptive enrichment design, clinical trial. Eligible patients with spontaneous BGH ≥20 mL will be randomized 1:1 to either minimally invasive endoscopic SCUBA evacuation plus standard medical management or standard medical management alone; the time of randomization will be used to classify participants in one of two cohorts: 1) those randomized <8 hours from onset, and 2) those randomized 8-16 hours from onset. Randomization is targeted to occur within 120 min of arrival to the randomizing center's Emergency Department (ED), and initiation of surgery is targeted to occur within 120 min of randomization. Participants will be followed at 30, 90, 180, and 365 days to assess for adverse events (AEs) and utility-weighted modified Rankin Scale (UW-mRS).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 80 years
* Non-traumatic, spontaneous, supratentorial, non-thalamic, BGH of volume ≥ 20 mL, as determined by the treating physician using ABC/2 method
* NIHSS ≥ 6 at presentation
* Computed Tomography Angiography (CTA) or Magnetic Resonance Angiography (MRA) is performed and does not show an underlying vascular lesion
* Pre-ICH mRS 0-2 Informed consent from patient or legally authorized representative (LAR) to participate in the trial, wherein patient/LAR's stated wishes are to pursue lifesaving therapies as opposed to early withdrawal of care (explicitly explained as <7 days following ictus)
* The treating physician anticipates that surgery can be initiated <120 min from randomization
* Randomization can occur ≤16 hours from LKW

Exclusion Criteria:

* Suspected secondary cause for the ICH, such as an underlying vascular malformation (cavernous malformation, arteriovenous malformation, etc.), aneurysm, neoplasm, hemorrhagic transformation of an underlying ischemic infarct; or venous infarct Infratentorial or thalamic hemorrhage
* Midbrain extension/involvement
* Coagulopathy defined as international normalized ratio (INR) > 1.4
* Elevated activated Partial Thromboplastin Time (aPTT) > 40 s
* Concurrent use of direct oral anticoagulants or low molecular weight heparin at ICH onset
* Known hereditary or acquired hemorrhagic diathesis or coagulation factor deficiency
* Platelet count <100 x 103 cells/mm3, or known platelet dysfunction (reversal of coagulopathy is not allowed) GCS score <7 at presentation
* Evidence of active infection indicated by fever ≥100.7 °F and/or open draining wound at the time of enrollment
* Any comorbid disease or condition expected to compromise survival or ability to complete follow-up assessments through 365 days
* Intraventricular extension of the hemorrhage is visually estimated to involve > 50% of either of the lateral ventricles
* Pregnancy (women of childbearing potential must have a negative pregnancy test to participate)
* Based on investigator's judgment, the patient does not have the necessary mental capacity to participate or is unwilling to comply with the protocol follow-up schedule
* Current participation in another interventional (drug or device) trial
* Pre-existing Do Not Resuscitate (DNR)/Do Not Intubate (DNI) status
* History of severe dementia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2030-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Utility-Weighted Modified Rankin Scale (UW-mRS) | Day 180
  Utility-Weighted Modified Rankin Scale (UW-mRS), a tool used primarily in stroke research to measure a patient's disability. It assigns a "utility" value (representing quality of life) to each level of the standard Modified Rankin Scale (mRS) to provide a more nuanced, patient-centered outcome measure than the mRS alone.
  The utility weighted mRS scales the 0-6 mRS range onto a 0-1 range, with higher scores indicating better health outcomes.

SECONDARY OUTCOMES:
Number of successful endoscopic clot removal | during procedure
  Successful endoscopic clot removal to ≤10 mL remaining clot
Volume of clot remaining post endoscopic clot removal | 24 hours post procedure
  Volume of clot remaining on follow-up 24-hour CT scan post endoscopic clot removal
Number of post-procedural complications adverse events | up to 30 days
  Symptomatic rebleeding into the cavitary lesion after evacuation resulting in residual hematoma volume >10 mL and worsening of neurological status (defined as an increase in pre-evacuation NIHSS ≥4 points or a decrease in GCS ≥2 points which cannot be attributed to any other cause such as infection, seizures, sedation, or worsening edema) within 30 days.
Number of CNS infection | Day 30
  CNS infection attributed to surgery
Mortality (all-cause) | Day 30
  Number of mortalities, for any reason, at day 30

CONTACTS AND LOCATIONS:
Overall Officials: J Mocco, MD, Principal Investigator — Mount Sinai Hospital System; Magdy Selim, MD, PhD, Principal Investigator — Harvard Medical School (HMS and HSDM); Sharon Yeatts, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Mount Sinai Health System, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Will follow StrokeNet and NIH data sharing guidelines
Access Criteria: Submission of (and subsequent approval of) request for use to the appropriate repository.